CLINICAL TRIAL: NCT06275763
Title: Optimal Medical Treatment of Difficult-to-treat Hypertension
Acronym: OPTIMAL-HT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/ABM/01/00037
Record Dates: First submitted 2024-01-04; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Eplerenone; Spironolactone; Torsemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Eplerenone (+placebo of Spironolactone and placebo of Torasemide) (Experimental): Phase C. Participants randomly assigned to this arm take Eplerenone and placebos of Spironolactone and Torasemide
  Interventions: Drug: Phase C: Eplerenone; Drug: Phase B: Triplixam / Elestar HCT
- Spironolactone (+placebo of Eplerenone and placebo of Torasemide) (Experimental): Phase C. Participants randomly assigned to this arm take Spironolactone and placebos of Eplerenone and Torasemide
  Interventions: Drug: Phase C: Spironolactone; Drug: Phase B: Triplixam / Elestar HCT
- Torasemide (+placebo of Eplerenone and placebo of Spironolactone ) (Experimental): Phase C. Participants randomly assigned to this arm take Torasemide and placebos of Eplerenone and Spironolactone
  Interventions: Drug: Phase C: Torasemide; Drug: Phase B: Triplixam / Elestar HCT
- Open-label (Active Comparator): Phase B Replacement of ineffective antihypertensive treatment based on 3 or more antihypertensive drugs (single or dual drug preparations) with a triple single pill combination (SPC) based on optimally combined antihypertensive drugs: perindopril + indapamide + amlodipine (P+I+A) or olmesartan + hydrocholothiazide + amlodipine (O+H+A).
  Interventions: Drug: Phase B: Triplixam / Elestar HCT
- Screening (Other): Phase A. Confirmation of the true ineffectiveness of antihypertensive therapy based on 3 or more antihypertensive drugs (single or dual drug preparations) using ABPM and home BP measurements.
  Interventions: Diagnostic Test: Phase A: Confirmation of uncontrolled hypertension

INTERVENTIONS:
Drug: Phase C: Eplerenone — Participants randomly assigned to this arm take Eplerenone and placebos of Spironolactone and Torasemide
  Other Names: Eplerenone
  Arms: Eplerenone (+placebo of Spironolactone and placebo of Torasemide)
Drug: Phase C: Spironolactone — Participants randomly assigned to this arm take Spironolactone and placebos of Eplerenone and Torasemide
  Other Names: Spironolactone
  Arms: Spironolactone (+placebo of Eplerenone and placebo of Torasemide)
Drug: Phase C: Torasemide — Participants randomly assigned to this arm take Torasemide and placebos of Eplerenone and Spironolactone
  Other Names: Torasemide
  Arms: Torasemide (+placebo of Eplerenone and placebo of Spironolactone )
Drug: Phase B: Triplixam / Elestar HCT — Replacement of ineffective antihypertensive treatment based on 3 or more antihypertensive drugs (single or dual drug preparations) with a triple single pill combination (SPC) based on optimally combined antihypertensive drugs: perindopril + indapamide + amlodipine (P+I+A) or olmesartan + hydrocholothiazide + amlodipine (O+H+A).
  Other Names: Triple Single Pill Combination: Triplixam / Elestar HCT
  Arms: Eplerenone (+placebo of Spironolactone and placebo of Torasemide); Open-label; Spironolactone (+placebo of Eplerenone and placebo of Torasemide); Torasemide (+placebo of Eplerenone and placebo of Spironolactone )
Diagnostic Test: Phase A: Confirmation of uncontrolled hypertension — Confirmation of the true ineffectiveness of antihypertensive therapy based on 3 or more antihypertensive drugs (single or dual drug preparations) using ABPM and home BP measurements.
  Arms: Screening

SUMMARY:
The purpose of this study is to evaluate best medical management to achieve the BP goals of ESC/ESH (120-129 / 70-79 mmHg) in HT patients who are <65 years old and ineffectively treated (BP ≥ 130/80 mg) with 3 or more antihypertensive drugs

DETAILED DESCRIPTION:
Purpose: To evaluate best medical management to achieve the ESC/ESH 2018 BP goals of 120-129 / 70-79 mmHg in HT patients aged < 65 y not controlled on 3 or more antihypertensive drugs.

Study design:

Phase A (Active screening) (n = 2500) 7 days Confirmation of the true ineffectiveness of antihypertensive therapy based on 3 or more antihypertensive drugs (single or dual drug preparations) using ABPM and home BP measurements.

Phase B (Open-label, non-randomized) (n = 1250) 12 weeks Replacement of ineffective antihypertensive treatment based on 3 or more antihypertensive drugs (single or dual drug preparations) with a triple single pill combination (SPC) based on optimally combined antihypertensive drugs: perindopril + indapamide + amlodipine (P+I+A) or olmesartan + hydrocholothiazide + amlodipine (O+H+A).

Phase C (Double blind, randomized, parallel-group) (n = 480) 24 weeks

Comparison of antihypertensive efficacy and tolerability profile:

* spironolactone
* eplerenone
* torasemide attached as an antihypertensive drug of 4th choice.

ELIGIBILITY:
Inclusion Criteria:

* documented history of HT
* HT treated for at least six months,
* office BP ≥ 130 and / or ≥80 mm Hg (average seated BP at Visit 1)
* use of 3 or more antihypertensive drugs, including an ACEi/ARB and a thiazide/thiazide-like diuretic or loop diuretic (single drugs or double SPCs)
* stable antihypertensive treatment regimen - no changes in antihypertensive treatment strategy at least for 4 weeks
* able and willing to comply with all study procedures and able to attend one of the study centers

Exclusion Criteria:

* inability to give informed consent
* SBP ≥180 mm Hg and/or DBP ≥110 mm Hg and/or DBP <60 mm Hg
* BMI ≥40 kg/m2
* eGFR of <45 mL/min/1.73 m2
* potassium serum concentration > 4.8 mmol/L or < 3.5 mmol/L
* persistent hyponatremia or history of hyponatremia related to TD/TLD treatment (sodium concentration <135 mmol/L)
* secondary hypertension (not including sleep apnea)
* chronic oral glucocorticoid therapy
* myocardial infarction or cerebrovascular event (e.g. stroke, transient ischemic event, cerebrovascular accident) in the year prior to study inclusion
* heart failure requiring treatment with diuretic or aldosterone antagonists
* cardiomyopathy exluding LVH related to HT
* severe valvular disease
* ascending aortic aneurysm ≥5 cm
* prescribed to any standard antihypertensive of cardiovascular medication (e.g. beta blockers) for other chronic conditions (e.g. chronic coronary syndromes, arytmia) such that discontinuation might pose serious risk to health
* primary pulmonary hypertension
* decompensated hyperthyroidism or hypothyroidism
* severe liver dysfunction (alanine aminotransferase and/or asparagine aminotransferase activity ≥3 times the upper limit of normal value),
* documented contraindication or allergy to studied drugs
* limited life expectancy of < 1 year at the discretion of the Investigator
* any known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or for any reason in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements
* all women of child bearing potential; women of child bearing potential can be included in the study ONLY after providing documentation of effective contraception (intrauterine device);
* concurrent enrollment in any other investigational drug or device trial
* anticipated change of medical status during the trial (e.g., surgical intervention requiring >2 weeks convalescence)
* current therapy for cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients with uncontrolled BP on ABPM | First week of the patients' participation in the study
  Percentage of patients with uncontrolled BP confirmed on ABPM (24h mean, SBP ≥125 mm Hg or DBP ≥80 mm Hg)
Patients with controlled BP after 12 weeks on triple SPC | Next 12 weeks of the patients' participation in the study
  Percentage of patients with controlled BP after 12 weeks of treatment with triple SPC, confirmed on ABPM (24h mean, SBP <125 mm Hg and DBP <80 mm Hg) - as the efficacy of the treatment strategy (switching ineffective treatment to triple SPC) - the whole group and P+I+A and E+H+A groups separetly.
Systolic BP reduction on 4th antihypertensive drug | Last 24 weeks of the patients' participation in the study
  Magnitude of reduction of SBP on ABPM (24h mean) after 12 weeks of treatment - comparison of eplerenone vs spironolactone and torasemide vs spironolactone.

SECONDARY OUTCOMES:
Percentage of patients with BP controlled confirmed by HBPM | First week of the patients' participation in the study
  Percentage of patients with BP controlled confirmed by HBPM (mean over the period of 6 days, SBP ≥130 mm Hg or DBP ≥80 mm Hg)
Consistency of the rate of uncontrolled BP | First week of the patients' participation in the study
  Consistency of the rate of uncontrolled BP between ABPM and HBPM
Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by OBPM | Next 12 weeks of the patients' participation in the study
  Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by OBPM (SBP <130 mm Hg and DBP <80 mm Hg).
Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by HBPM | Next 12 weeks of the patients' participation in the study
  Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by HBPM (mean over 6 days, SBP <130 mm Hg and DBP <80 mm Hg).
Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by ABPM | Next 12 weeks of the patients' participation in the study
  Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by ABPM in daytime (SBP <135 mm Hg and DBP <85 mm Hg) and nighttime (SBP <120 mm Hg and DBP <70 mm Hg) reading.
Percentage of patients requiring an increase in the dose | Next 12 weeks of the patients' participation in the study
  Percentage of patients requiring an increase in the dose of drugs used in the whole group and in the patients treated with P+I+A and O+H+A separately.
Consistency of the rate of uncontrolled BP | Next 12 weeks of the patients' participation in the study
  Consistency of the rate of uncontrolled BP between ABPM, HBPM and OBPM.
The magnitude of the decrease in SBP and DBP on OBPM, ABPM and HBPM after 12 weeks | Next 12 weeks of the patients' participation in the study
  The magnitude of the decrease in SBP and DBP on OBPM, ABPM and HBPM after 12 weeks of treatment in the whole group and in the patients treated with P+I+A and O+H+A separately.
The magnitude of changes in HBPM and ABPM derived indices after 12 weeks | Next 12 weeks of the patients' participation in the study
  The magnitude of changes in HBPM and ABPM derived indices after 12 weeks of treatment in the whole group and in the patients treated with P+I+A and O+H+A separately.
Phase C | Last 24 weeks of the patients' participation in the study
  * Changes of SBP on ABPM (24h mean) after 12 weeks of treatment in patients receiving spironolactone, eplerenone or torasemide as compared against baseline.
  * Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by OBPM (SBP <130 mm Hg and DBP <80 mm Hg) - comparison of eplerenone / torasemide groups against the spironolactone group.
  * Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by HBPM (mean over 6 days, SBP <130 mm Hg and DBP <80 mm Hg) - comparison of eplerenone / torasemide groups against the spironolactone group.
  * Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by ABPM, in 24h mean (SBP <125 mm Hg and DBP <80 mm Hg), daytime (SBP <135 mm Hg and DBP <85 mm Hg) and nighttime (SBP <120 mm Hg and DBP <70 mm Hg) readings - comparison of eplerenone / torasemide groups against the spironolactone group.
Changes of SBP on ABPM (24h mean) after 12 weeks of treatment | Last 24 weeks of the patients' participation in the study
  Changes of SBP on ABPM (24h mean) after 12 weeks of treatment in patients receiving spironolactone, eplerenone or torasemide as compared against baseline.
Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by OBPM | Last 24 weeks of the patients' participation in the study
  Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by OBPM (SBP <130 mm Hg and DBP <80 mm Hg) - comparison of eplerenone / torasemide groups against the spironolactone group.
Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by HBPM | Last 24 weeks of the patients' participation in the study
  Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by HBPM (mean over 6 days, SBP <130 mm Hg and DBP <80 mm Hg) - comparison of eplerenone / torasemide groups against the spironolactone group.
Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by ABPM | Last 24 weeks of the patients' participation in the study
  Percentage of patients with controlled BP after 12 weeks of treatment, confirmed by ABPM, in 24h mean (SBP <125 mm Hg and DBP <80 mm Hg), daytime (SBP <135 mm Hg and DBP <85 mm Hg) and nighttime (SBP <120 mm Hg and DBP <70 mm Hg) readings - comparison of eplerenone / torasemide groups against the spironolactone group.
Phase C continuation | Last 24 weeks of the patients' participation in the study
  Consistency of the rate of controlled BP between ABPM, HBPM and OBPM (after 12 weeks of treatment).
Phase C continuation | Last 24 weeks of the patients' participation in the study
  Changes in SBP and DBP on OBPM, ABPM and HBPM after 12 weeks of treatment - comparison of eplerenone / torasemide groups against the spironolactone group and comparison of each of the studied drug groups against baseline.
Changes in HBPM and ABPM derived indices after 12 weeks - comparison of treatment groups | Last 24 weeks of the patients' participation in the study
  Changes in HBPM and ABPM derived indices after 12 weeks of treatment - comparison of eplerenone / torasemide groups against the spironolactone group and comparison of each of the studied drug groups against baseline
Changes of SBP on ABPM (24h mean) after 24 weeks of treatment compared against spironolactone | Last 24 weeks of the patients' participation in the study
  Changes of SBP on ABPM (24h mean) after 24 weeks of treatment in patients receiving eplerenone or torasemide as compared against spironolactone.
Changes of SBP on ABPM (24h mean) after 24 weeks of treatment compared against baseline | Last 24 weeks of the patients' participation in the study
  Changes of SBP on ABPM (24h mean) after 24 weeks of treatment in patients receiving spironolactone, eplerenone or torasemide as compared against baseline.
Percentage of patients with controlled BP after 24 weeks of treatment, confirmed by OBPM - comparison between groups | Last 24 weeks of the patients' participation in the study
  Percentage of patients with controlled BP after 24 weeks of treatment, confirmed by OBPM (SBP <130 mm Hg and DBP <80 mm Hg) - comparison of eplerenone / torasemide groups against the spironolactone group.
Percentage of patients with controlled BP after 24 weeks of treatment, confirmed by HBPM - comparison between groups | Last 24 weeks of the patients' participation in the study
  Percentage of patients with controlled BP after 24 weeks of treatment, confirmed by HBPM (mean over 6 days, SBP <130 mm Hg and DBP <80 mm Hg) - comparison of eplerenone / torasemide groups against the spironolactone group.
Percentage of patients with controlled BP after 24 weeks of treatment, confirmed by ABPM - comparison between groups | Last 24 weeks of the patients' participation in the study
  Percentage of patients with controlled BP after 24 weeks of treatment, confirmed by ABPM, in 24h mean (SBP <125 mm Hg and DBP <80 mm Hg), daytime (SBP <135 mm Hg and DBP <85 mm Hg) and nighttime (SBP <120 mm Hg and DBP <70 mm Hg) readings - comparison of eplerenone / torasemide groups against the spironolactone group.
Consistency of the rate of controlled BP between ABPM, HBPM and OBPM after 24 weeks | Last 24 weeks of the patients' participation in the study
  Consistency of the rate of controlled BP between ABPM, HBPM and OBPM after 24 weeks of treatment
Changes in SBP and DBP on OBPM, ABPM and HBPM after 24 weeks of treatment - comparison between groups | Last 24 weeks of the patients' participation in the study
  Changes in SBP and DBP on OBPM, ABPM and HBPM after 24 weeks of treatment - comparison of eplerenone / torasemide groups against the spironolactone group and comparison of each of the studied drug groups against baseline.
Changes in HBPM and ABPM derived indices after 24 weeks of treatment - - comparison between groups | Last 24 weeks of the patients' participation in the study
  Changes in HBPM and ABPM derived indices after 24 weeks of treatment - comparison of eplerenone / torasemide groups against the spironolactone group and comparison of each of the studied drug groups against baseline
Percentage of patients requiring an increase in the dose of drugs used after 6 and 12 weeks - comparison between groups | Last 24 weeks of the patients' participation in the study
  Percentage of patients requiring an increase in the dose of drugs used after 6 and 12 weeks - comparison of eplerenone / torasemide groups against the spironolactone.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Dobrowolski, Professor, Principal Investigator — National Institute of Cardiology
Locations (1):
- National Institute of Cardiology, Warsaw, Masovian Voivodeship, Poland